CLINICAL TRIAL: NCT04815525
Title: The Longterm Risk of Advanced Colorectal Neoplasia After Colonoscopy - A Population-based Cohort Study in Hong Kong
Acronym: ACNC
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Resident Specialist, Chinese University of Hong Kong
Other Study IDs: 2020.597
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Neoplasia; Colorectal Cancer
Keywords: colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal finding: Colonoscopy finding normal
- Hyperplastic polyps: Colonoscopy finding of hyperplastic polyps
- Low-risk adenomas: Colonoscopy finding of low-risk adenomas
- High-risk adenomas: Colonoscopy finding of high-risk adenomas

SUMMARY:
The primary objective of this study is to analyze the 15-year cumulative incidence of advanced colorectal neoplasia and CRC-related mortality after the index colonoscopy.

DETAILED DESCRIPTION:
This is a territory-wide retrospective observational cohort study using the Clinical Data Analysis and Reporting System (CDARS). We will identify patients from CDARS with colonoscopy performed from 1 January 2000 to 31 October 2020. Other relevant diagnoses, procedures, concomitant drugs, laboratory parameters and pathology results will be retrieved and studied.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with colonoscopy performed in HA hospitals during the study period would be eligible for screening.

Exclusion Criteria:

1. Patients with documented personal history of colorectal cancers before the study period would be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will identify patients from CDARS with colonoscopy performed from 1 January 2000 to 31 October 2020. Other relevant diagnoses, procedures, concomitant drugs, laboratory parameters and pathology results will be retrieved and studied.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Culumative incidence of advanced colorectal neoplasia | 15 years
  high-risk adenomas or CRC after 15 years of index conoloscopy

SECONDARY OUTCOMES:
CRC-related mortality rate | 15 years
  the rate of mortality due to CRC-related incidents

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD with other researchers